CLINICAL TRIAL: NCT01877486
Title: Pulmonary Vein Isolation Using Cryoablation Alone in Paroxysmal Atrial Fibrillation Patients Converted From Persistent Atrial Fibrillation With Dofetilide
Brief Title: PVI Using Cryoablation Alone in Paroxysmal AF Patients Converted From Persistent AF With Dofetilide
Acronym: ABLATE
Status: Withdrawn | Type: Observational
Why Stopped: funding not available
Sponsor: University of Rochester (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Jonathan S. Steinberg, Adjunct Professor of Medicine, University of Rochester
Other Study IDs: UR Cryo PVI
Record Dates: First submitted 2013-05-26; First posted 2013-06-13 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
Keywords: atrial fibrillation; cryoballoon ablation; persistent AF; paroxysmal AF; dofetilide
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cryoballoon ablation: After pre-treatment with dofetilide and conversion of persistent AF to sinus rhythm, performance of PVI using cryoballoon
  Interventions: Procedure: Ablation

INTERVENTIONS:
Procedure: Ablation — Pulmonary vein isolation following dofetilide

SUMMARY:
To determine the efficacy of cryoablation alone in patients with paroxysmal atrial fibrillation who have been pretreated with dofetilide and converted from persistent atrial fibrillation.

DETAILED DESCRIPTION:
Pulmonary vein isolation is now considered a cornerstone of all atrial fibrillation (AF) ablation procedures. In patients with paroxysmal AF, pulmonary vein isolation alone is usually sufficient. The cryoballoon is now FDA approved to achieve PVI in patients with paroxysmal AF.

Although no ablation system is yet approved in patients with persistent AF, these patients are increasingly undergoing ablation. Many investigators feel that these patients have more atrial disease and thus PVI alone is insufficient in these patients. As a result, it is common for these patients to undergo additional ablation, which is often quite extensive and exposes patients to proarrhythmia. Commonly utilized strategies include linear lesions (left atrial roof; mitral isthmus line), ablation of complex fractionated atrial electrograms (CFAEs), left atrial appendage isolation and/or even right atrial ablation. For years, the investigators have been concerned about the adverse effects of this additional ablation. The investigators postulated that the "answer" is not more ablation but trying to "reverse remodel" patients with persistent AF back to a paroxysmal form, whereby PVI alone would again be justified and sufficient. The efficacy of such a strategy has previously been demonstrated.

In brief, the investigators start patients with persistent AF on dofetilide 3 months prior to scheduled ablation. In 96% of patients, AF either suppresses completely or is transformed into a paroxysmal pattern. The net effect is "reverse remodeling" of the left atria. The investigators have confirmed this by using a reduction in P wave duration as a surrogate of remodeling. At the ablation procedure, the investigators perform PVI alone.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years
* Able and willing to give written informed consent
* Paroxysmal AF, defined as recurrent AF ( ≥ 2 episodes in 1 month) that terminates within 7 days as assessed by ECG recordings
* Prior persistent AF, defined as sustained beyond seven days and up to one year, successfully converted to paroxysmal AF by dofetilide

Exclusion Criteria:

* Previous ablation for AF
* Left atrial size larger than 60mm (parasternal view on transthoracic echocardiogram)
* Patients who have AF episodes triggered by another uniform arrhythmia (e.g. atrial flutter or atrial tachycardia)
* Presence of severe valvular disease with the need for surgical correction
* AF deemed secondary to a transient or correctable abnormality including electrolyte imbalance, trauma, recent surgery, infection, toxic ingestion, and endocrinopathy
* Pregnant women or women of child bearing potential and not on reliable methods of birth control
* Second or third degree AV block, sinus pause > 3 seconds, resting heart rate< 30 bpm without permanent pacemaker
* History of drug-induced Torsades de Pointes or congenital long QT syndrome
* Uninterrupted AF for more than 12 months prior to randomization unless sinus rhythm maintained for ≥ 24 hours after cardioversion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for catheter ablation of AF
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation/flutter | One year
  As assessed by one week Holters and symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Steinberg, MD, Principal Investigator — University of Rochester
Locations (1):
- Valley Hospital, Ridgewood, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No